CLINICAL TRIAL: NCT03136315
Title: Renal Function Evaluation in an Ultra Endurance Race: On the Interest of Monitoring Specific Biomarkers to Asses Renal Risk.
Brief Title: Evaluation of the Renal Function in an Ultra-endurance Race.
Acronym: INFERNAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017-A00808-45
Record Dates: First submitted 2017-04-21; First posted 2017-05-02 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-04

CONDITIONS: Renal Insufficiency, Acute
Keywords: Renal failure; athlete; ultra endurance
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- INFERNAL Arm (Experimental): The INFERNAL Arm will have serum and urinary dosage for creatinine and cystanin C at the beginning and at the end of the 110 km race.
  Interventions: Other: INFERNAL Intervention

INTERVENTIONS:
Other: INFERNAL Intervention — The intervention consists in serum and urinary dosage (creatinine and Cystatin C) at the beginning and the end of the 110 km race.

SUMMARY:
During ultra endurance events, athletes experience extreme physical and mental demands, sometimes at the limits of the adaptive response to human physiology. This is particularly true for the renal function, and some evidence for acute renal failure has already been shown, sometimes leading to dialysis. However, the precise mechanisms involved in acute renal failure in such ultra endurance races are not clearly elucidated.

The aim of our study is to estimate glomerular filtration rate from serum and urinary creatinine and cystitin C at the beginning and at the end of a 110 km ultra endurance race. Our hypothesis is that during the ultra endurance race, renal function may be injured, with a risk for the athlete.

ELIGIBILITY:
Inclusion Criteria:

* Age: At least 20 years old
* Athlete that is officially registered to the 110 km race (INFERNAL Trail des Vosges)
* Athlete informed by a member (MD) of the Medical Staff of the race.
* Athlete that gives and signes the informed consent to the research protocol

Exclusion Criteria:

* Athlete with a known disease that needs the following medications:
* Medications influencing the renin-angiotensin-aldosteron system (angiotensin-converting enzyme inhibitors, angiotensin receptor blockers, aldosteron receptor blockers)
* Diuretic drugs
* Anticoagulant drugs
* Non-steroidal anti-inflammatory drugs
* Athlete with a known thyroid disease (because of the influence on the serum cystatin level)
* Athlete with a know renal disease
* Athlete with a know inflammatory disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2017-09-10 (Actual); Study Completion 2017-09-10 (Actual)

PRIMARY OUTCOMES:
Glomerular filtration rate | 30 minutes at baseline (09.07.2017), and 30 minutes at the end of the 110 km race (2 or 3 days after baseline)
  The glomerular filtration rate will be calculated from the serum and urinary creatinine and cystatin C dosage

CONTACTS AND LOCATIONS:
Locations (1):
- Stade des Perrey, Saint-Nabord, Lorraine, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Didier S, Vauthier JC, Gambier N, Renaud P, Chenuel B, Poussel M. Substance use and misuse in a mountain ultramarathon: new insight into ultrarunners population? Res Sports Med. 2017 Apr-Jun;25(2):244-251. doi: 10.1080/15438627.2017.1282356. Epub 2017 Jan 23. PMID 28114830
- [Background] Poussel M, Vauthier JC, Renaud P, Gambier N, Chenuel B, Ladriere M. [Acute kidney injury following naproxene use in an ultraendurance female athlete]. Presse Med. 2013 Sep;42(9 Pt 1):1274-6. doi: 10.1016/j.lpm.2012.09.030. Epub 2013 Feb 27. No abstract available. French. PMID 23453505
- [Background] Hoffman MD, Weiss RH. Does Acute Kidney Injury From an Ultramarathon Increase the Risk for Greater Subsequent Injury? Clin J Sport Med. 2016 Sep;26(5):417-22. doi: 10.1097/JSM.0000000000000277. PMID 26657822
- [Background] Hoffman MD, Stuempfle KJ, Fogard K, Hew-Butler T, Winger J, Weiss RH. Urine dipstick analysis for identification of runners susceptible to acute kidney injury following an ultramarathon. J Sports Sci. 2013;31(1):20-31. doi: 10.1080/02640414.2012.720705. Epub 2012 Oct 4. PMID 23035796